CLINICAL TRIAL: NCT03025698
Title: A Phase II, Open-label, Non-controlled, Intra-patient Dose-escalation Study to Characterize the Pharmacokinetics After Oral Administration of Eltrombopag in Pediatric Patients With Refractory, Relapsed or Treatment Naive Severe Aplastic Anemia or Recurrent Aplastic Anemia
Brief Title: A Phase II Dose-escalation Study Characterizing the PK of Eltrombopag in Pediatric Patients With Previously Untreated or Relapsed Severe Aplastic Anemia or Recurrent Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CETB115E2201
Record Dates: First submitted 2017-01-12; First posted 2017-01-19 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Aplastic Anemia
Keywords: Eltrombopag; Horse anti-thymocyte globulin; Cyclosporine; previously untreated or relapsed severe aplastic anemia; recurrent aplastic anemia; Severe aplastic anemia; Pharmacokinetics; Immunosuppressive therapy; ETB115; Refractory
MeSH Terms: conditions — Anemia, Aplastic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Option 1) (Experimental): Regimen 1: hATG (ATGAM®), CsA and eltrombopag begin on Day 1.
  Interventions: Drug: Eltrombopag; Drug: hATG; Drug: CsA
- Cohort A (option 2) (Experimental): CsA and eltrombopag begin on Day 1.
  Interventions: Drug: Eltrombopag; Drug: CsA
- Cohort B (Experimental): previously untreated SAA, hATG (ATGAM®), CsA and eltrombopag begin on Day 1 and all patients will be treated with the same regimen
  Interventions: Drug: Eltrombopag; Drug: hATG; Drug: CsA

INTERVENTIONS:
Drug: Eltrombopag — Tablet for oral use, once daily or Powder for oral suspension (PfOS), once daily
  Other Names: ETB115
Drug: hATG — Horse ATG (ATGAM) (hATG) is not considered an investigational medicinal product (IMP)
  Arms: Cohort A (Option 1); Cohort B
Drug: CsA — Cyclosporine (CsA) will be by supplied as either oral capsules or oral solution, administered twice a day

SUMMARY:
This is a phase II, open label, multi-center, intra-patient dose escalation study to characterize the pharmacokinetics (PK) after oral administration of eltrombopag in combination with immunosuppressive therapy in pediatric patients with previously untreated or relapsed/refractory severe aplastic anemia or recurrent aplastic anemia.

DETAILED DESCRIPTION:
All patients were treated with eltrombopag for the 26-week Treatment Period, followed by a 52-week Follow-Up Period. Patients who had been previously untreated with immunosuppressive therapy were treated according to the standard of care, hATG/cyclosporine, in addition to eltrombopag. Patients with relapsed/refractory SAA or recurrent AA were enrolled into one of two treatment options: hATG/cyclosporine plus eltrombopag or cyclosporine plus eltrombopag, depending on prior treatment with immunosuppressive therapy. Patients could receive eltrombopag beyond 26 weeks if the investigator thought that the patient was still receiving clinical benefit from the drug.

After initiating treatment with eltrombopag, patients had their dose assessed and modified as tolerated, until the targeted platelet count or maximum dose was achieved. Pharmacokinetic assessments were performed at time points intended to capture steady state PK of the starting dose and highest dose achieved.

There are four separate periods of this study: Screening (signing of written informed consent through Day -1), Treatment (for 26 weeks), Follow-up (additional 52 weeks), and Long-term Follow-up (for additional 3 years). The first 3 periods were considered the Core phase of the study.

Study completion (Core) will occur when the last patient completes the 26-week treatment and 52-week Follow-up Period [at Week 78].

ELIGIBILITY:
Inclusion Criteria:

For Cohort A patients:

* History of prior diagnosis of SAA,
* Diagnosis of relapsed/refractory SAA or recurrent AA following treatment for SAA, as per Section 5.1. Patients with recurrent AA (e.g., losing their response) are exempt from meeting the diagnostic criteria for SAA relapse at the time of study enrollment, but must have been previously diagnosed with SAA.
* Agree to concurrent eltrombopag treatment with appropriate, investigator-selected Immunosuppressive therapy (IST) with either hATG + CsA or CsA.

For Cohort B patients:

* Diagnosis of SAA at time of enrollment.
* Patients must not have been previously treated with IST, and must meet all criteria as described in Table 5-1.
* Patients must agree to treatment with hATG + CsA concurrent with eltrombopag.

All patients eligible for inclusion in this study must meet all of the following criteria:

* Age 1 to <18 years.
* Assessments to rule out congenital/inherited bone marrow failure syndromes and other causes of immune-mediated pancytopenia, which may be treated with transplant, must be completed prior to enrollment.
* Hematopoietic stem cell transplantation (HSCT) is not suitable or available as a treatment option or has been refused by the patient. (Candidacy for HSCT will be determined as per local practices or national guidelines.)
* Bone marrow aspirate and biopsy at any time during the 4 weeks prior to first dose of eltrombopag.
* Performance status score: Karnofsky ≥50 for patients 16 years of age and older or Lansky ≥50 for patients below 16 years of age.
* Written informed consent must be signed by a parent or legal guardian prior to initiation of any study specific procedure.
* Normal karyotype within 4 weeks prior to first dose of eltrombopag. If there are insufficient metaphases (< 10) to determine karyotype, a repeat marrow aspirate is required. If upon repeat bone marrow aspirate, the number of metaphases is insufficient (< 10), then FISH probes performed in marrow aspirate as per protocol must be normal.

Exclusion Criteria:

* Prior and/or active medical history of:

  * Fanconi anemia (via chromosome breakage test or growth arrest by flow cytometry)
  * Other known underlying inherited marrow failure syndrome (such as but not limited to Dyskeratosis Congenita, Congenital Amegakaryocytic Thrombocytopenia, or Shwachman-Diamond Syndrome).
* Symptomatic Paroxysmal Nocturnal Hemoglobinuria (PNH) and/or PNH clones >50% of White blood cell (WBC) or Red blood cell (RBC) at time of enrollment.

  * Any cytogenetic abnormalities by karyotyping or FISH.
  * Myelodysplastic syndrome (MDS)
  * Other known or suspected underlying primary immunodeficiency
  * Any malignancy
* Active infection not responding to appropriate therapy.
* Prior eltrombopag or other thrombopoietin receptor (TPO-R) agonist treatment for at least 2 months and a lack of response.
* Have any of the following out-of-range laboratory values:

  * Serum Creatinine >2.5 × upper limit of normal (ULN),
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 × ULN.
* Concurrent participation in an investigational study within 30 days prior to enrollment or within 5-half-lives of the investigational product, whichever is longer. Note: a parallel enrollment in a registry for patients with SAA or AA is acceptable.

Pregnant or nursing (lactating) women.

* Female patients of childbearing potential (e.g., are menstruating or could reach menarche during the study, this usually includes girls 9 years and older) who do not agree to abstinence or, if sexually active, do not agree to the use of contraception as defined in Section 7.2.1.2.6 (pregnancy section) of the protocol. If local regulations are more stringent than the contraception methods listed in this protocol to prevent pregnancy, local regulations apply and will be described in the ICF.
* Male patients who are sexually active and do not agree to abstinence or to use a condom during intercourse while taking eltrombopag, and for 13 weeks after stopping treatment.
* Patients, who in the investigators' opinion may be unwilling, are unable or unlikely to comply with the requirements of the study protocol.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to eltrombopag or its excipient, CSA, or hATG that contraindicates patient participation.
* History of major surgery, serious illness, or traumatic injury within 4 weeks of first dose of study treatment.
* Patients with known history of HIV positivity.
* Patients with known history of hepatitis B or C positivity.
* Any severe and/or uncontrolled medical conditions which could cause unacceptable safety risks or compromise compliance with the protocol, such as:

  • Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome),Active skin, mucosa, ocular or GI disorders of Grade > 1.
* Impaired cardiac function, such as:

  * Patients with a history of congenital long QT syndrome or known family history of long QTc syndrome,
  * Corrected QTc >450 msec using Fridericia correction (QTcF) on the screening ECG (using triplicate ECGs),
  * Ventricular arrhythmias and or other cardiac arrhythmia not controlled with medication,
  * Other clinically significant cardio-vascular disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension),
  * History of known structural abnormalities (e.g., cardiomyopathy).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Eltrombopag PK parameter: AUCtau | at the highest dose level, i.e. 11 weeks after dose initiation
  Area under the curve calculated to the end of the dosing interval (tau).
Eltrombopag PK parameter: Cmax | at the highest dose level, i.e. 11 weeks after dose initiation
  Peak concentration of drug
Eltrombopag PK parameter: Ctrough | at the highest dose level, i.e. 11 weeks after dose initiation
  Pre-dose drug concentration in a repeated dose setting.

SECONDARY OUTCOMES:
Percentage of participants who have achieved a complete (CR) or partial response (PR) | Week 12, Week 26, Week 52, and Week 78.
  Percentage of participants who have achieved a complete (CR) or partial response (PR)
Percentage of participants with a platelet response | Week 12, Week 26, Week 52, and Week 78.
  Percentage of participants who have achieved a complete or partial platelet response
Hematologic counts | Week 12, Week 26, Week 52, Week 78, and then annually up to 3 years
  Platelet (PLT), Hgb, and neutrophil counts
Red Blood Cell (RBC) transfusion independence | From date of first dose to approx. 3 years
  Number and frequency of participants with RBC transfusion independence defined as a period of time of at least 56 days without RBC transfusion.
Platelet transfusion independence | From date of first dose to approx. 3 years
  Number and frequency of participants with platelet transfusion independence defined as a period of time of at least 28 days without PLT transfusion.
Bone marrow cellularity | Screening, Week 12, Week, 26, Week 52, Week 78 and then annually up to 3 years
  Percentage of hematopoietic cells in bone marrow biopsy.
Bone marrow morphology | Screening, Week 12, Week, 26, Week 52, Week 78 and then annually up to 3 years
  Percentage of hematopoietic cells in bone marrow aspirate
Bone marrow cytogenetics | Screening, Week 12, Week, 26, Week 52, Week 78 and then annually up to 3 years
  Chromosomal structure by karyotyping and Fluorescence in situ hybridization (FISH)
Acceptability and palatability for both tablets and powder for oral suspension | Week 1, Week 2, Week 3, Week 4, Week, 12, Week 26, Week 78
  Standardized (total) summary score, ranged from 0-100 will be derived from all items from the questionnaire based on a scoring matrix.
Clonal evolution to Paroxysmal Nocturnal Hemoglobinuria (PNH) | Baseline, Week 12, 26, 52, 78 and annually for up to 3 years to at time of disease progression.
  Percentage of participants with PNH clones
Exposure-response relationship of eltrombopag and overall response and platelet response | Week 12 or up to Week 26 when the PK highest dose has been achieved
  Pharmacokinetic parameters of eltrombopag at the highest dose by the best overall response and platelet response
Alternate Overall response (aOR) | Week 12, Week 26, Week 52, and Week 78.
  Percentage of participants with alternate overall response rate (aORR) defined as the proportion of patients who have achieved an alternate complete response (aCR) or an alternate partial response (aPR)
PK of eltrombopag at the starting dose (AUCtau) | Week 3 Day 1
  Pharmacokinetic parameters of eltrombopag (AUCtau)
PK of eltrombopag at the starting dose (Cmax) | Week 3 Day 1
  Pharmacokinetic parameters of eltrombopag (Cmax)
PK of eltrombopag at the starting dose (Ctrough) | Week 3 Day 1
  Pharmacokinetic parameters of eltrombopag (Ctrough)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (12):
  - Phoenix Children s Hospital, Phoenix, Arizona
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - Childrens Hospital Colorado, Aurora, Colorado
  - Aflac Cancerand Blood Disorders Ctr, Atlanta, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Childrens Hosp Boston Dept of Hematology, Boston, Massachusetts
  - University of MI Health System, Ann Arbor, Michigan
  - Hackensack University Medical Center SC-2, Hackensack, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Texas Children's Cancer and Hematology Center, Houston, Texas
- Novartis Investigative Site, Shatin, Hong Kong
- Novartis Investigative Site, Lisbon, Portugal
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Thailand (2):
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shimamura A, Maschan A, Bennett C, Samarasinghe S, Farrar JE, Li CK, Sirachainan N, Pongtanakul B, Komvilaisak P, Zubarovskaya L, Rothman JA, Walkovich K, Nakano TA, Bertuch AA, Ferrao A, Bhat R, Hanna R, Overholt K, Boklan J, Wong TF, Wang Q, Urban P, Strahm B, Wang W, Vlachos A, Williams DA. Eltrombopag in combination with immunosuppressive therapy in pediatric severe aplastic anemia: phase 2 ESCALATE trial. Blood Adv. 2025 Aug 12;9(15):3728-3738. doi: 10.1182/bloodadvances.2024015102. PMID 40315366